CLINICAL TRIAL: NCT01277653
Title: Prospective, Randomized Study of PIVKA-II and AFP Measurement Every 3 Months Compared to AFP Every 6 Months in Surveillance Program for Early Detection of Hepatocellular Carcinoma
Brief Title: Study of PIVKA-II and AFP Measurement in Surveillance Program for Early Detection of Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Collaborators: Severance Hospital (Other)
Responsible Party: Do Young Kim, Department of Internal Medicine, Yonsei University College of Medicine
Other Study IDs: AFP-PIVKA
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2011-01-17 (Estimated); Status verified 2009-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- PIVKA-II and AFP 6 months: PIVKA-II and AFP measurement every 6 months
- tumor maker interval every 6 month: tumor maker interval every 6 month
  Interventions: Device: tumor maker interval shortly

INTERVENTIONS:
Device: tumor maker interval shortly — tumor maker interval every 3 month
  Other Names: tumor maker interval every 3 month
  Groups: tumor maker interval every 6 month

SUMMARY:
There is no prospective study on the test intervals of alpha-fetoprotein (AFP) or on the role of prothrombin induced vitamin K absence or antagonist-II (PIVKA-II) in surveillance program for early detection of hepatocellular carcinoma(HCC). The goal of this study is to compare if the testing of AFP + PIVKA-II in intervals of 3 months is more effective in diagnosing early stages of HCC than the 6 month interval of AFP that is commonly used

DETAILED DESCRIPTION:
There is no prospective study on the test intervals of alpha-fetoprotein (AFP) or on the role of prothrombin induced vitamin K absence or antagonist-II (PIVKA-II) in surveillance program for early detection of hepatocellular carcinoma(HCC). The goal of this study is to compare if the testing of AFP + PIVKA-II in intervals of 3 months is more effective in diagnosing early stages of HCC than the 6 month interval of AFP that is commonly used

ELIGIBILITY:
Inclusion Criteria:

* LC

Exclusion Criteria:

* previous HCC

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver cirrhosis
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2007-06; Primary Completion 2010-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
the difference of curative treatments & survival rates | 4 years

SECONDARY OUTCOMES:
the difference of early detection rates of HCC between both groups | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Myoung HA LEE, MD, Study Director — OFF
Locations (1):
- Severance Hospital, Seoul, Seodaemun-gu, South Korea